CLINICAL TRIAL: NCT04822441
Title: Prospective Study on the Risks of Dengue Fever for the Fetus.
Acronym: ERiDenF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/CHU/14
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-03

CONDITIONS: Dengue Fever
Keywords: dengue fever ; pregnancy
MeSH Terms: conditions — Dengue | interventions — Data Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients who contracted dengue fever before 34 weeks of amenorrhea: Patients who contracted biologically proven dengue fever during pregnancy before 34 weeks outside the peri-partum period (more than 12 days before childbirth)
  Interventions: Other: data collection
- Patients who contracted dengue fever after 34 weeks of amenorrhea: Patients who contracted biologically proven dengue fever during pregnancy after 34 weeks outside the peri-partum period (more than 12 days before childbirth)
  Interventions: Other: data collection
- Patients who have contracted dengue during the peripartum period: Patients who have contracted dengue during the peripartum period or who have a suspicion of dengue (in the 12 days preceding childbirth)
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — Ultrasound follow-up maternal dengue serology PCR (Polymerase Chain Reaction) and dengue serology of the umbilical cord

SUMMARY:
Dengue is the most common arbovirus worldwide (390 million people infected each year) and belongs to the Flavivirus genus of the Flaviviridae family like Zika. Its expansion has been rapid since the last decade with an increase in the number of cases of 400% and the first cases of indigenous dengue described in Europe.

Current data on the consequences of dengue fever on the fetus are incomplete. The risk of maternal-fetal transmission of dengue during the peripartum period has now been recorded in numerous case reports and a few case series for patients who contracted dengue in the 12 days preceding childbirth or at the time of delivery. However, the transmission of dengue is highly variable depending on the studies ranging from 1.6 to 15% and the consequences for the newborn are very variable ranging from simple thrombocytopenia to death in severe neonatal dengue.

Regarding the risk of malformation, a few old cases of heart disease, hydrocephalus and neural tube closure abnormalities have been described in the literature following exposure to dengue fever during pregnancy. Since no malformative case has been described, however, to our knowledge, no prospective study with specialized ultrasound monitoring has been performed for pregnant women who contracted dengue during their pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients
* Major
* Affiliated with social security
* Symptomatic or pauci-symptomatic dengue
* Biological confirmation of dengue fever by dengue positive PCR or IgM positive during the current dengue episode

Exclusion Criteria:

* Multiple pregnancy
* Patient's refusal
* Protected persons: person deprived of liberty by judicial or administrative decision, minor, and person subject to a legal protection measure: guardianship or curators)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who contracted dengue fever during pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-03-19 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Study the teratogenic effects of the dengue virus on the fetus | at childbirth
  Rate of fetal anomalies such as infectious fetal disease or any other fetal anomaly detected during specialized antenatal ultrasound follow-up.

SECONDARY OUTCOMES:
Study the maternal-fetal transmission of dengue fever during pregnancy | at childbirth
  Amniotic fluid positive dengue PCR (Polymerase Chain Reaction) rate
Study the maternal-fetal transmission of dengue fever in the peri-partum | at childbirth
  Umbilical cord dengue positive and / or IgM (immunoglobulin M) positive PCR rate
Study the materno-placental transmission of dengue fever during pregnancy and peri-partum | at childbirth
  Placental dengue positive PCR rate
Study the consequences at the placental level of dengue, in terms of anatomopathological alterations | at childbirth
  Placental pathology abnormalities rate

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de la Réunion, Saint-Pierre, France

IPD SHARING:
Plan to Share IPD: No